CLINICAL TRIAL: NCT02596503
Title: A Phase I/II Study of Eribulin in Combination With Oral Irinotecan for Adolescent and Young Adult Patients With Relapsed or Refractory Solid Tumors
Brief Title: A Study of Eribulin in Combination With Oral Irinotecan for Adolescent and Young Adult Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0659.cc; NCT02318589 (obsolete NCT alias)
Record Dates: First submitted 2015-10-19; First posted 2015-11-04 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Relapsed Solid Tumors; Refractory Solid Tumors
Keywords: young adults; adolescents
MeSH Terms: interventions — eribulin; Irinotecan; Cefixime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eribulin + Irinotecan (Experimental): Eribulin will be administered intravenously on days 1 and 8 of a 21-day cycle, while irinotecan will be administered orally on days 1-5. The oral antibiotic cefixime will be used to reduce irinotecan-associated diarrhea.
  Eribulin dose will be assigned at time of enrollment using a 3+ 3 Phase 1 design (ranging from 0.8 - 1.4 mg/m2/dos). The dose of irinotecan will be fixed at 90 mg/m2/day x 5 days.
  Interventions: Drug: Eribulin; Drug: Irinotecan; Other: Cefixime

INTERVENTIONS:
Drug: Eribulin — Intravenous eribulin administered on days 1 and 8 of a 21-day cycle.
Drug: Irinotecan — Irinotecan will be administered orally at a fixed dose of 90 mg/m2/day on days 1 -5 of a 21-day cycle.
Other: Cefixime — Cefixime will be given to all patients to reduce irinotecan-associated diarrhea. It will be administered Day -1 through Day 8 of each cycle.
  Other Names: Suprax

SUMMARY:
This IND-exempt Phase I trial will establish the recommended Phase II (RP2D) dose of eribulin in combination with fixed doses of oral irinotecan in adolescents and young adults with relapsed or refractory solid tumors. Eribulin will be administered intravenously on days 1 and 8 of a 21-day cycle, while irinotecan will be administered orally on days 1-5.

Patients will be assigned an eribulin dose level at the time of enrollment using a 3+3 Phase I design, and there will be no intrapatient dose escalation. Once the RP2D has been established, there will be up to 10 patients enrolled in a dose expansion cohort. In absence of disease progression or toxicity, subjects may receive up to 17 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must ≥13 and ≤30 years of age at the time of study entry
* Patients must have a histologically confirmed solid tumor malignancy at either original diagnosis or relapse for which no curative therapy exists, and which has either recurred or progressed after at least one prior systemic therapy. Patients with primary brain tumors, or those with brain metastases at time of potential enrollment, are excluded. Additionally, patients with GIST, alveolar soft part sarcoma, or dematofibrosarcoma protuberans are excluded.
* Patients must have either measurable or evaluable disease,
* Performance Level: ECOG performance status ≤ 2 (Karnofsky ≥60%, see Appendix A). Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purposes of assessing the performance score.
* Prior Therapy: No limit is placed on the number of prior therapies. Prior treatment with irinotecan or eribulin is allowed, although patients must not have received co-administration of eribulin and irinotecan and must not have had disease progression while receiving either eribulin or irinotecan.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  * Myelosuppressive chemotherapy: Must not have received within three weeks of start date of this protocol chemotherapy; six weeks is required after administration of nitrosourea agents.
  * Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor or at least 14 days for a long-acting growth factor (e.g. pegfilgrastim)
  * Biologic (anti-neoplastic agent): At least 7 days or 3 half-lives since the completion of therapy with a biologic agent, whichever is longer. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are expected to occur. The duration of this interval must be discussed with the PI of the study.
  * Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy (e.g. tumor vaccines).
  * Monoclonal antibodies: At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody.
  * Radiotherapy: ≥ 2 weeks for local palliative XRT (small port); ≥ 6 months must have elapsed if prior TBI, craniospinal XRT; ≥ 3 months must have elapsed if ≥ 50% radiation of pelvis; ≥ 6 weeks must have elapsed if therapeutic doses of MIBG or other substantial BM irradiation was given.
  * Stem Cell Transplant or Rescue without TBI: Allogeneic and autologous HSCT will be allowed, if there is no evidence of active graft vs. host disease and ≥ 2 months must have elapsed since infusion. Patients must not be on systemic immunosuppression.
* Organ Function Requirements: Patients must have normal organ and marrow function as defined below.
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 100,000/mcL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
* Hemoglobin ≥ 8.0 g/dl (may receive RBC transfusions).
* Total bilirubin ≤ 1.5 × institutional upper limit of normal for age
* AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal
* Albumin ≥ 2 g/dl
* Creatinine within normal institutional limits for age OR creatinine clearance ≥ 70 mL/min/1.73 m2 for patients with creatinine levels above normal
* EKG QTc ≤480 msec (CTCAE Grade 2)
* Contraception: Because chemotherapeutic agents may be teratogenic, males and females of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 4 months after the last dose of study chemotherapy.
* Informed Consent: All patients > 18 years must sign a written informed consent. Patients < 18 years old must provide assent, and the parent or legal guardian must sign the written informed consent.

Exclusion Criteria:

* Pregnancy or Breast-Feeding: Patients who are pregnant or breast-feeding are not eligible for this study due to the potential for fetal or teratogenic toxicities. Negative pregnancy tests must be obtained in female patients who are post-menarchal.
* Major surgery within 14 days prior to start of treatment. No time limitations after minor surgery (eg: core biopsy or central line placement)
* Current evidence of GIST, alveolar soft part sarcoma, or dermatofibrosarcoma
* Concomitant Medications:

  * Growth factor(s): Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment (14 days if pegfilgrastim).
  * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible.
  * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
  * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
  * Enzyme-inducing anticonvulsants or other medications: Patients who are currently receiving the enzyme inducing anticonvulsants: phenytoin, phenobarbital, carbamazepine, oxcarbazepine are not eligible. Patients who are currently taking rifampin, voriconazole, itraconazole, ketoconazole, aprepitant, or St. John's Wort are not eligible.
  * Anticoagulants: Use of warfarin is not allowed while on study. Patients already on warfarin should use alternative anticoagulants while on this study. Warfarin must not have been administered within 7 days of starting protocol therapy.
  * Medications that prolong the QTc:
* Infection: Patients who have an uncontrolled infection, or who are currently receiving treatment for C difficile infection.
* Patients with a history of allergic reactions attributed to eribulin or irinotecan.
* Patients with documented allergy to cephalosporins.
* Patients with CNS tumors or known brain metastases.
* Patients with known metastatic tumor in the bone marrow.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with eribulin and irinotecan. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
The recommended Phase II dose of eribulin when used in combination with oral irinotecan | Within 2 years
  To estimate the recommended phase II dose of eribulin in combination with fixed-dose oral irinotecan in adolescents and young adults with relapsed/refractory solid tumors. A 3+3 trial design will be utilized. Accrual will continued based on DLT evaluation until the RP2D is established and at least 6 patients have been treated at this dose.

SECONDARY OUTCOMES:
The number of patients with adverse events (according to CTCAE V.4) in patients receiving the combination of eribulin and irinotecan | Within 2 years
  The intensity of AEs will be graded according to the CTCAE V.4 on a 5-point scale
The best overall response based on RECIST 1.1 criteria | Within 2 years
  To estimate the anti-tumor effects of the eribulin and irinotecan drug combination using RECIST 1.1 criteria
The area under the plasma concentration versus time curve of eribulin in adolescent and young adult patients receiving oral irinotecan | 2 years
  Pharmacokinetic measurements will be performed on days 1 and 8 of the first cycle
The peak plasma clearance, Cmax, of eribulin in adolescent and young adult patients receiving oral irinotecan | 2 years
  Pharmacokinetic measurements will be performed on Days 1 and 8 of the first cycle
The half-life of eribulin in adolescent and young adults patients receiving oral irinotecan | 2 years
  Pharmacokinetic measurements will be performed on Days 1 and 8 of the first cycle

CONTACTS AND LOCATIONS:
Overall Officials: Carrye Cost, MD, Principal Investigator — University of Colorado, Denver; Tom Badgett, MD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Kentucky, Lexington, Kentucky
  - University of Texas, Southwestern Medical Center, Dallas, Texas

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT02596503/Prot_SAP_ICF_000.pdf